CLINICAL TRIAL: NCT00194727
Title: Weekly Vinorelbine and Oral Capecitabine as Treatment for Stage IV Breast Cancer: A Phase II Trial With Molecular Correlates
Brief Title: Weekly Vinorelbine and Oral Capecitabine as Treatment for Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Hoffmann-La Roche (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20912-A; 02-1544-A 06 (Other: UW Human Subjects Division)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Breast Neoplasm
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Vinorelbine (20 mg/m2 IV weeks 1, 2 and 3 of each 3 week cycle) and capecitabine (825 mg/m2 twice a day; days 1 - 14 of each 3 week cycle). Treatment continues until disease progression, excessive toxicity or other reason to remove patient from protocol therapy.
  Interventions: Drug: Vinorelbine; Drug: Capecitabine

INTERVENTIONS:
Drug: Vinorelbine — 20 mg/m2 IV weeks 1, 2 and 3 of each 3 week cycle. Treatment continues until disease progression, excessive toxicity or other reason to remove patient from protocol therapy.
Drug: Capecitabine — 825 mg/m2 twice a day; days 1 - 14 of each 3 week cycle. Treatment continues until disease progression, excessive toxicity or other reason to remove patient from protocol therapy.

SUMMARY:
The primary purpose of the study is to examine the safety and effectiveness of combination therapy consisting of daily oral capecitabine and weekly intravenous vinorelbine in stage IV breast cancer subjects. The study is designed to assess the safety and effectiveness of this combination therapy. Safety will be assessed by analyzing the types of toxicity, the severity of toxicity and the need for dose modification or delay due to toxicity. Effectiveness will be assessed by analyzing response rates, time to treatment failure, time to progression and overall survival. Our hypothesis is that the regimen will be more effective than standard historic regimens for this type and stage of cancer.

DETAILED DESCRIPTION:
Single-agent chemotherapy is rarely curative in advanced breast cancer. Combination regimens are the next logical step in the attempt to improve tumor response rates and prolong survival. Oral capecitabine is a convenient way to deliver drug a 5-fluorouracil analogue. In addition, vinorelbine is a newer vinca alkaloid chemotherapeutic agent with improved efficacy and probably improved toxicity over its predecessors in the treatment of breast cancer. We propose combining these two agents. As these two drugs have non-overlapping toxicities and differing mechanisms of action, we anticipate being able to deliver both drugs in near full dose.

Secondary purposes include assessing whether there is a correlation between intra-tumoral enzyme levels and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be older than 18 and younger than 85.
* Subject must have metastatic (stage IV) breast cancer.
* Subject must have pathologic confirmation of breast cancer (at least of primary disease). Biopsy confirmation of stage IV disease is desirable but not required. Tissue blocks must be available for review.
* Subject must have measurable or non-measurable disease as defined below:

Measurable disease includes lesions that can be accurately measured in at least one dimension as greater than 2.0 cm with conventional techniques or as greater than 1.0 cm with spiral CT scan.

Non-measurable disease includes all other lesions (e.g. lesions less than 2.0 cm by conventional techniques or less than 1.0 cm by spiral CT, bone lesions, pleural effusion, etc.).

- Subject must be willing and able to provide informed consent.

Exclusion Criteria:

* Subject must not have significant co-morbid conditions such as clinically significant cardiac disease not well controlled with medication (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias), or myocardial infarction within the last 12 months or serious concurrent infection.
* Subject must not have rapidly progressing visceral involvement (e.g. liver, lymphangitic lung).
* Subject must not have evidence of CNS metastases.
* Subject must not have abnormal hematologic values (neutrophils less than 1.5 x 103/uL, platelet count less than 100 x 103/uL).
* Subject must not have impaired renal function (serum creatinine greater than 1.5 x upper normal limit) or estimated creatinine clearance below 30 mL/min by the Cockcroft and Gault equation.
* Subject must not have serum bilirubin greater than 1.5 x upper normal limit.
* Subject must not have ALT or AST greater than 2.5 x upper normal limit (or greater than 5 x upper normal limit in the case of liver metastases).
* Subject must not have alkaline phosphatase greater than 2.5 x upper normal limit (or greater than 5 x upper normal limit in the case of liver metastases or greater than 10 x upper normal limit in the case of bone disease).
* Subject must not have a lack of physical integrity of the upper gastrointestinal tract, inability to swallow or malabsorption syndrome
* Subject must not have a history of fluoropyrimidine therapy (unless given in an adjuvant setting and completed at least 12 months earlier).
* Subject must not have a life expectancy less than 3 months.
* Subject must not have a Karnofsky Performance Status less than 70%.
* Subject must not have a history of another carcinoma within the last five years except non-melanoma skin and treated in-situ cervical cancer.
* Subject must not have a history of unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil.
* Subject must not have organ allografts.
* Subject must not be pregnant or lactating woman. (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential).
* Subject must not be less than four weeks from completion of previous chemotherapy regimen or with related toxicities unresolved prior to the start of study treatment.
* Subject must not be less than four weeks from major surgery or without complete recovery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Best response as determined at the time that the subject completes protocol treatment | <= 4 years

SECONDARY OUTCOMES:
Time to progression as determined at the time that each subject's disease worsens following treatment | <= 4 years
Median survival at two and three years following the start of protocol treatment. | <= 3 years
Correlation between intra-tumoral enzyme levels and prognosis | <= 4 years
Measure the toxicity of the regimen | During study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Georgiana K. Ellis, M.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington; Seattle Cancer Care Alliance, Seattle, Washington, United States